CLINICAL TRIAL: NCT04793061
Title: Circulating Tumor DNA as Marker for Response to Antineoplastic Treatment of Metastatic Cancer (FLUIDO)
Acronym: FLUIDO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Elisabethinen Hospital (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Holger Rumpold, Head GI-Cancer Center, Elisabethinen Hospital
Other Study IDs: FLUIDO-001
Record Dates: First submitted 2021-03-09; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Cancer
Keywords: metastatic cancer, circulating tumor DNA, treatment, response prediction
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for isolation of cell free DNA for the detection of circulating tumor specific DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sample collection — Blood is samples from peripheral vein during routine care

SUMMARY:
Early monitoring of antineoplastic treatment benefit is a central medical need. Radiologic assessment for documentation of response is done after several months of treatment usually. This implies that patients not responding are exposed to unnecessary toxicity. According to several reports showing the correlation of the amount of circulating tumour DNA with tumour burden we aim to investigate its early dynamic change at the beginning and during antineoplastic treament until radiologic response assessment. Blood samples necessary for that are taken within the scope of clinical routine care. We hypothesize that the changes of circulating tumour DNA correlate with the radiological findings.

DETAILED DESCRIPTION:
Patients Patients with metastatic cancer who are treated with antineoplastic treatment are eligible if a molecular marker is either known due to the type of cancer (Case A) or if a molecular marker is known due to routine assessment (Case B). An example for "Case A" is pancreatic cancer, which is known to harbor KRAS-mutations as part of tumorigenesis in more than 90% (8), or multiple cancers harboring methylated WIF(9). A typical example for "Case B" is colorectal or gastric cancer. Systemic treatment requires the knowledge of the mutational status of RAS, EGFR and BRAF, which is assessed routinely from tumor tissue. If a mutation is found the patient qualifies for participation in the project. We finally plan to include at least 40 patients with mPDAC, another 40 patients with mCRC and 20 patients with mGC (100 patients in total at least).

* The inclusion criteria therefore are:

  * Metastatic cancer (mPDAC, mGC, mCRC)
  * Known mutation of the cancer
  * Signed informed consent
  * At least 18 years
  * Eligible for antineoplastic treatment
  * Patient treated at the Ordensklinikum Linz
* Exclusion criteria o Inclusion criteria not met

Treatment monitoring Circulating tumor DNA is analysed from peripheral blood. For this purpose, 30 ml blood is taken at start and during treatment additionally to the blood volume required for analyses in the frame of routine. Therefore, there are no extra blood sampling time points additionally to these required for routine care. Due to that, the time points depend on the cancer type investigated as treatment schedules are different. However, within an entity the time points are homogenous.

Analysis of ctDNA The preparation of ctDNA is done in the Laboratory for Molecular Biology and Tumor Cytogenetics at the Ordensklinikum Linz (Dr. Gerald Webersinke) and digital droplet PCR is performed by the Department of Genetics at the Medical University of Innsbruck (Prof. Johannes Zschoke). The analysis is performed in a batch and not in real time. In detail, ctDNA detection is based on KRAS-screening in mPDAC or by patient specific ddPCR. The latter patient specific ddPCR is based on the mutations found in the tumor by NGS-screening (ARCHER or Truesight 170 or whole-genome sequencing if panels are negative) at the Laboratory in Linz. This is the case for mGC and mCRC, where multiple mutations are possible (KRAS, NRAS, BRAF, TP53). In patients suffering from mCRC, this analysis in performed within routine procedures as such mutations are crucial for treatment decisions. In case of mGC mutations screening is done within the proposed project.

Radiology assessment Assessment of treatment response is performed as part of the routine treatment after two to three months of treatment at the department of Radiology of the Ordensklinikum Linz.

Statistics Data are analyzed in order to detect a dependency between ctDNA dynamics and response to treatment. Method for example is chi-square test. Software used is RStudio Version 1.2.5019.

Descriptive Statistics Mean, standard deviation, minimum and maximum for every concentration of ctDNA at each time point.

ROC-AUC analysis for every time point

* Dynamics of ctDNA concentration at every time point (metric variable)
* Outcome after 12 weeks as a dichotome variable (responder [SD/PR/CR], non-responder)
* Calculation of AUC with 95% CI (all time points)
* ROC-curve (all time points)
* Calculation of sensitivity and specificity for all time points with 95% CI
* Determination of the optimal threshold-value upon sensitivity and specificity for every time point
* Comparison of predictive value of each time point based on sensitivity/specificity, AUC by CI-values

Power-analysis Based on the current patient recruitment we assume to end up with a final number of 100 patients.

Assumptions:

* n = 100
* Power 80 %
* Significance-niveau 5 %, Confidence-Intervall (CI) 95 %
* Proportion of responders (estimated prevalence): 0.2, 0.4 and 0.6
* Sensitivity and specificity: 0.6, 0.7 and 0.8
* Dropout-rate: 15 %

Plan for analysis We first compare Roc curves at the different timepoints to identify the timepoint that as the best tradeoff between performance and gain of time (lack of power to provide statistical comparisons). In a second step, we identify the best cut point of ctDNA at the chosen timepoint based on youden index for instance and give sensitivity/specitivity and also NPV/PPV at this cut-point.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic cancer (mPDAC, mGC, mCRC)
* Known mutation of the cancer
* Signed informed consent
* At least 18 years
* Eligible for antineoplastic treatment

Exclusion Criteria:

o Inclusion criteria not met

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic cancer who are treated with antineoplastic treatment are eligible if a molecular marker is either known due to the type of cancer (Case A) or if a molecular marker is known due to routine assessment (Case B). An example for "Case A" is pancreatic cancer, which is known to harbor KRAS-mutations as part of tumorigenesis in more than 90% (8), or multiple cancers harboring methylated WIF(9). A typical example for "Case B" is colorectal or gastric cancer. Systemic treatment requires the knowledge of the mutational status of RAS, EGFR and BRAF, which is assessed routinely from tumor tissue. If a mutation is found the patient qualifies for participation in the project. We finally plan to include at least 40 patients with mPDAC, another 40 patients with mCRC and 20 patients with mGC (100 patients in total at least).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
ctDNA dynamics correlate with response to antineoplastic treatment | 3 months per patient
  ctDNA concentration in peripheral blood will drop if patient respond to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ordensklinikum Linz, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No